CLINICAL TRIAL: NCT00907998
Title: A Randomized, Double-blind, Placebo-controlled, Multiple Dose Study in Patients With Coronary Heart Disease (CHD) to Assess Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Subcutaneous Administration of APL180
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of APL180
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CAPL180A2210B; EudraCT 2009-010877-19
Record Dates: First submitted 2009-05-22; First posted 2009-05-25 (Estimated); Last update posted 2009-11-20 (Estimated); Status verified 2009-11

CONDITIONS: Coronary Heart Disease
Keywords: Coronary heart disease; APL180
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- APL180 (first dose level) (Experimental)
  Interventions: Drug: APL180
- APL180 (second dose level) (Experimental)
  Interventions: Drug: APL180
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: APL180
  Arms: APL180 (first dose level)
Drug: APL180
  Arms: APL180 (second dose level)
Drug: Placebo
  Arms: Placebo

SUMMARY:
The design of this study will enable an extensive evaluation of safety, tolerability, and PK-PD relationship following 4 weeks of dosing in patients with Coronary heart Disease

ELIGIBILITY:
Inclusion Criteria:

* Male and female CHD or CHD equivalent patients
* Body mass index (BMI) must be within the range of 20 to 35 kg/m2,
* Patient must have been on a stable statin therapy for >8 weeks prior to first dose except for the statin intolerant patients.

Exclusion criteria:

* Pregnancy
* Significant illness within two weeks prior to dosing.
* Triglycerides ≥ 500 mg/dl (5.65 mmol/l)
* Uncontrolled hypertension
* Any condition that in the opinion of the investigator or the Novartis medical monitor would jeopardize the evaluation of efficacy or safety.
* Presence of NYHA Class III or IV chronic heart failure
* MI or angioplasty (including stenting), acute coronary syndrome (ACS), unstable angina or arterial embolic disease within 6 months prior to do Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2009-06; Primary Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of APL180 | Throughout the study

SECONDARY OUTCOMES:
Pharmacokinetics of APL180 | Throughout the study
Evaluate effects of APL180 biomarkers | Throughout the study
Pharmacokinetic-pharmacodynamic relationship of APL180 | Throughout the study
Effect of APL180 on exploratory biomarkers, | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (11):
- United States (3):
  - Pinnacle Research Group, Anniston, Alabama
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Icon Clinical Research, San Antonio, Texas
- Novartis Investigator Site, Copenhagen, Denmark
- Germany (3):
  - Novartis Investigator Site, Mainz
  - Novartis Investigator Site, Mannheim
  - Novartis Investigator Site, Neuss
- Israel (3):
  - Novartis Investigator Site, Rehovot
  - Novartis Investigator Site, Tel Aviv
  - Novartis Investigator Site, Zrifin
- Novartis Investigator Site, Amsterdam, Netherlands